CLINICAL TRIAL: NCT04936945
Title: Comparative Study Between the Outcome of Intra-articular Injection of Platelet Rich Plasma Versus Hyaluronic Acid in Arthroscopic Management of Temporomandibular Degenerative Joint Diseases: A Randomized Clinical Trial
Brief Title: Intra-articular Injection in Arthroscopic Management of Temporomandibular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd-elmoniem, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-21-06-15
Record Dates: First submitted 2021-06-13; First posted 2021-06-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthroscopy plus platelet rich plasma. (Active Comparator): Group A: will be treated with operative arthroscopy plus intra-articular injection of platelet rich plasma
  Interventions: Procedure: Temporomandibular joint arthroscopy plus intra-articular injection
- arthroscopy plus hyaluronic acid. (Active Comparator): Group B: will be treated with operative arthroscopy plus intra-articular injection of hyaluronic acid
  Interventions: Procedure: Temporomandibular joint arthroscopy plus intra-articular injection

INTERVENTIONS:
Procedure: Temporomandibular joint arthroscopy plus intra-articular injection — patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative diagnostic arthroscopic treatment then at the end of the procedure intra-articular injection of platelet rich plasma or hyaluronic acid will be done.

SUMMARY:
The aim of this study is to evaluate the efficacy of intra-articular injection of platelet rich plasma versus hyaluronic acid following diagnostic arthroscopy in the management of patients suffering from degenerative temporomandibular joint (TMJ).

This is a prospective randomized study of 20 patients with TMJ degenerative joint diseases Wilkes IV, V.

Patients will be divided into two groups; Group A: will be treated with operative arthroscopy plus intra-articular platelet rich plasma.

Group B: will be treated with operative arthroscopy plus intra-articular hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

* - All patients with reduced mouth opening and/or painful maximum mouth opening.
* Joint pain.
* Patients with radiological evidence of degenerative joint disease.
* Patients with unsuccessful medical conservative treatment for at least two months.
* Unilateral or bilateral temporomandibular joint involvement.
* Wilkes stages IV and V

Exclusion Criteria:

* - Patients with bony ankylosis .
* Patients with advanced resorption of the glenoid fossa.
* Patients with infection or tumors around joint area
* Patients unfit for intervention medically.
* Patients who refused to share in the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samia M Saied, MD, Study Chair — Professor
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arthroscopy Plus Platelet Rich Plasma.: Group A: will be treated with operative arthroscopy plus intra-articular injection of platelet rich plasma
  Temporomandibular joint arthroscopy plus intra-articular injection: patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative arthroscopic treatment then at the end of the procedure intra-articular injection of platelet rich plasma.
- Arthroscopy Plus Hyaluronic Acid.: Group B: will be treated with operative arthroscopy plus intra-articular injection of hyaluronic acid
  Temporomandibular joint arthroscopy plus intra-articular injection: patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative arthroscopic treatment then at the end of the procedure intra-articular injection of hyaluronic acid .
Period: Overall Study
Arm/Group | Arthroscopy Plus Platelet Rich Plasma. | Arthroscopy Plus Hyaluronic Acid.
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arthroscopy Plus Platelet Rich Plasma.: Group A: will be treated with operative arthroscopy plus intra-articular injection of platelet rich plasma
  Temporomandibular joint arthroscopy plus intra-articular injection: patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative diagnostic arthroscopic treatment then at the end of the procedure intra-articular injection of platelet rich plasma.
- Arthroscopy Plus Hyaluronic Acid.: Group B: will be treated with operative arthroscopy plus intra-articular injection of hyaluronic acid
  Temporomandibular joint arthroscopy plus intra-articular injection: patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative diagnostic arthroscopic treatment then at the end of the procedure intra-articular injection of hyaluronic acid.
- Total: Total of all reporting groups
Arm/Group | Arthroscopy Plus Platelet Rich Plasma. | Arthroscopy Plus Hyaluronic Acid. | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (9.94) | 31.9 (9.94) | 31.9 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Interincisal Opening (MIO) Measurements
Description: change in maximum inter-incisal mouth opening will be measured in millimeters between preoperative and postoperative at 1 week,3 weeks, the every month till 6 months
Time Frame: change from baseline maximum interincisal mouth opening in millimeters at 6 months postoperative
Measure: Mean (Standard Deviation); unit: Millimeter
Groups:
- Arthroscopy Plus Hyaluronic Acid.: Group B: will be treated with operative arthroscopy plus intra-articular injection of hyaluronic acid
  Temporomandibular joint arthroscopy plus intra-articular injection: patients with TMJ degenerative joint diseases Wilkes stages IV, V not responding to conservative treatment will undergo operative diagnostic arthroscopic treatment then at the end of the procedure intra-articular injection hyaluronic acid.
Arm/Group | Arthroscopy Plus Platelet Rich Plasma. | Arthroscopy Plus Hyaluronic Acid.
Number analyzed (Participants) | 10 | 10
Millimeter
  Pre-operative | 23.1 (6.71) | 27.9 (4.51)
  1-week PO | 33.8 (3.43) | 35.6 (3.96)
  3-weeks PO | 36 (4.4) | 36.7 (4.92)
  1-month PO | 36.7 (5.08) | 37.3 (5.5)
  2-months PO | 36.7 (5.08) | 37.6 (5.21)
  3-months PO | 37.6 (4.55) | 38.2 (4.71)
  4-months PO | 37.1 (4.41) | 38 (4.29)
  5-months PO | 36.8 (4.78) | 38.3 (4.06)
  6-months PO | 36.9 (4.95) | 38.5 (4.33)

2. Primary Outcome: Pain Intensity Measurements
Description: A 100 -point visual analogue scale (VAS) for the assessment of pain intensity with 0 as the absence of pain and 100 as the worst pain imaginable With filled standardized charts.
Time Frame: change from preoperative pain intensity according to 100 -point visual analogue scale at 6 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopy Plus Platelet Rich Plasma. | Arthroscopy Plus Hyaluronic Acid.
Number analyzed (Participants) | 10 | 10
score on a scale
  preoperative | 49 (20.79) | 49 (21.32)
  1-week PO | 28 (14.76) | 30 (14.14)
  3-weeks PO | 21 (8.76) | 25 (14.34)
  1-month PO | 16 (9.66) | 20 (14.91)
  2-months PO | 13 (6.75) | 13 (9.49)
  3-months PO | 12 (7.89) | 7 (4.83)
  4-months PO | 12 (10.33) | 4 (5.16)
  5-months PO | 14 (13.5) | 3 (4.83)
  6-months PO | 14 (13.5) | 3 (4.83)

ADVERSE EVENTS:
Time Frame: 23 months
Arm/Group | Arthroscopy Plus Platelet Rich Plasma. | Arthroscopy Plus Hyaluronic Acid.
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04936945/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04936945/SAP_001.pdf